CLINICAL TRIAL: NCT02522234
Title: A Phase Ib Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of F-627 as Prophylaxis Therapy to TAC Chemotherapy in Women With Breast Cancer
Brief Title: A Pharmacokinetics/Dynamics Ib Study of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Collaborators: Fudan University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-CDR-1-1301
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Neutropenia
Keywords: Neutropenia; Chemotherapy
MeSH Terms: conditions — Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- F-627 240 µg/kg (Experimental): F-627 at the dose of 240 mcg/kg administered by s.c. injection on Day 2 of each cycle for up to 6 cycles.
  Chemotherapy (docetaxol, doxorubicin and cyclophosphamide) administered by intravenous injection on Day 1 of each cycle for up to 6 cycles.
  Interventions: Biological: F-627 240 μg/kg
- F-627 320 µg/kg (Experimental): F-627 at the dose of 320 mcg/kg administered by s.c. injection on Day 2 of each cycle for 6 cycles.
  Chemotherapy (docetaxol, doxorubicin and cyclophosphamide) administered by intravenous injection on Day 1 of each cycle for up to 6 cycles.
  Interventions: Biological: F-627 320 μg/kg

INTERVENTIONS:
Biological: F-627 240 μg/kg — F-627 at 240 μg/kg dose enrolling 6 patients with breast cancer receiving adjuvant chemotherapy. Subjects will receive a corresponding dose of F-627 by subcutaneous injection 24 hours after each cycle（21 days） of chemotherapy drug administration. Blood samples are then collected at multiple time points during follow-up visits to evaluate the pharmacokinetics, pharmacodynamics, and safety of the drug. Dose will remain unchanged throughout the treatment period. Eligible subjects will be enrolled sequentially into the 240 μg/kg arm. And the arm should contain 6 evaluable subjects.
  Other Names: rh G-CSF Fc Fusion Protein
  Arms: F-627 240 µg/kg
Biological: F-627 320 μg/kg — F-627 at 320 μg/kg dose enrolling 6 patients with breast cancer receiving adjuvant chemotherapy. Subjects will receive a corresponding dose of F-627 by subcutaneous injection 24 hours after each cycle（21 days） of chemotherapy drug administration. Blood samples are then collected at multiple time points during follow-up visits to evaluate the pharmacokinetics, pharmacodynamics, and safety of the drug. Dose will remain unchanged throughout the treatment period. Eligible subjects will be enrolled sequentially into the 320 μg/kg arm. The arm should contain 6 evaluable subjects.
  Other Names: rh G-CSF Fc Fusion Protein
  Arms: F-627 320 µg/kg

SUMMARY:
This study was a phase Ib study of the safety and pharmacokinetics/pharmacodynamics of F-627 once per cycle as prophylaxis therapy to chemotherapy in women with breast cancer.

The patients received the intravenous administration of the chemotherapy (docetaxol, doxorubicin and cyclophosphamide, 75 mg/m2, 50 mg/m2 and 500 mg/m2 respectively) on Day 1 and the subcutaneous injection of F-627 at 240 µg/kg and 320 µg/kg on Day 2 (approximately 24 hours after chemotherapy) each cycle for up to 6 cycles.

DETAILED DESCRIPTION:
This study was a phase Ib study of the safety and pharmacokinetics/pharmacodynamics of F-627 once per cycle as prophylaxis therapy to chemotherapy in women with breast cancer.

This study was conducted at two centers in China and enrolled 15 patients with breast cancer receiving TAC chemotherapy (docetaxel, doxorubicin and cyclophosphamide). The patients received the intravenous administration of the chemotherapy (docetaxol, doxorubicin and cyclophosphamide, 75 mg/m2, 50 mg/m2 and 500 mg/m2 respectively) on Day 1 and the subcutaneous injection of F-627 at 240 µg/kg and 320 µg/kg on Day 2 (approximately 24 hours after chemotherapy) each cycle for up to 6 cycles. Patients will remain on study drug dose for each of the following 6 chemotherapy cycles.

Patients will remain on study drug dose for each of the following 6 chemotherapy cycles. The blood sampling will be collected for F-627 serum concentration analysis in cycle of 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. Female with breast cancer patients after resection who planned to receive up to 6 cycles of chemotherapy (docetaxol, doxorubicin and cyclophosphamide).
3. Score 0-1 of East Cooperative Oncology Group (ECOG).
4. Absolute neutrophil count (ANC) ≥ 2.0 × 109/L, hemoglobin (Hb) ≥ 11.0 g/dl, and platelets (PLT) ≥ 100 × 109/L prior to chemotherapy;
5. Liver and kidney function tests were within normal range;
6. Left ventricular ejection fraction (LVEF) > 50%;
7. Willing to provide written informed consent and to compliant study procedure.

Exclusion Criteria:

1. Pregnancy or lactating women; female with pregnancy potential had positive pregnancy test prior to study treatment.
2. Expected survival < 12 months.
3. Patients received radiotherapy within 4 weeks prior to enrollment.
4. Patients received neoadjuvant chemotherapy prior to the resection for breast cancer.
5. Patients received bone marrow or hemopoietic stem cell transplantation;
6. Patient was with malignancy other than breast cancer.
7. Patients received G-CSF treatment within 6 weeks prior to enrollment.
8. Patient cann't tolerate the pre-treatment of chemotherapy.
9. Acute congestive heart failure, myocardial disease, or myocardial infarction diagnosed by clinical, electrocardiography, or any other medical procedure.
10. Any disease that possibly cause splenomegaly.
11. Acute infections, chronic active hepatitis B infection within 1 year (except subject with negative hepatitis B antigen prior to enrollment) or history of hepatitis C infection.
12. Patients with active tuberculosis (TB), or had ever the history of close contact with patients with TB except negative result in tuberculin test; or under TB treatment; or suspected TB by chest X-ray.
13. Known the positive result of human immunodeficiency virus (HIV) or patients with acquired immune deficiency syndrome (AIDS).
14. Patients with sickle-cell anemia.
15. Patients with alcohol abuse or drug addiction that may affect the compliance of the study.
16. Patients with allergy to proteins extracted from Escherichia coli, G-CSF, or drug excipient.
17. Patients took other investigational products within 4 weeks prior enrollment.
18. Patients with diseases or symptoms that may not be suitable to be enrolled in this study based on investigator's judgment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2015-08-19 (Actual); Study Completion 2015-08-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events/abnormal laboratory value as measure of safety | Up to 6 cycles (about 126 days)
  Number of participants with adverse events/abnormal laboratory value as measure of safety and tolerability of rh G-CSF Fc fusion protein (F-627) in female patients wiht breast cance receiving adjuvant chemotherapy.

SECONDARY OUTCOMES:
Parameter of Peak Plasma Concentration | Cycle 1 and cycle 3 (each cycle was about 21 days)
  Parameter of Peak Plasma Concentration as a measure of pharmacokinetics profile of F-627.
Parameter of Area Under Plasma Concentration versus Time Curve | Cycle 1 and cycle 3 (each cycle was about 21 days)
  Parameter of Area Under Plasma Concentration versus Time Curve as a measure of pharmacokinetics profile of F-627.
Parameter of Clearance | Cycle 1 and cycle 3 (each cycle was about 21 days)
  Parameter of Clearance as a measure of pharmacokinetics profile of F-627.
Absolute Neutrophil Count changes over time | Up to 6 cycles (about 126 days)
  Absolute Neutrophil Count changes over time as measure of pharmacodynamics of F-627.

OTHER OUTCOMES:
Immunogenicity of F-627 | Up to 6 cycles (about 126 days)
  Immunogenicity of F-627 by serum anti-F-627 antibody analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, Professor, Principal Investigator — Fudan Universtiy Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China